CLINICAL TRIAL: NCT06069869
Title: Individually Randomized Crossover Trial of Multiple Micronutrient Supplementation (MMS) Iron Dosages During Pregnancy in Tanzania
Brief Title: Multiple Micronutrient Supplementation (MMS) Iron Dose Acceptability Crossover Trial
Acronym: MID-ACT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Ifakara Health Institute (Other); Harvard School of Public Health (HSPH) (Other); Muhimbili University of Health and Allied Sciences (Other); Africa Academy for Public Health (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Emily Smith, Principal Investigator, George Washington University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MID-ACT
Record Dates: First submitted 2023-09-15; First posted 2023-10-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Pregnancy Related
Keywords: Acceptability; Multiple Micronutrient Supplementation; Iron; Tanzania

STUDY DESIGN:
Intervention Model Description: Each participant will be randomized to one of 6 sequence orders to receive the three MMS regimens first, second or third in order (e.g., 30, 45, then 60 mg; or 45, 30, then 60 mg; or 45, 60 then 30 mg etc.).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial is quadruple blind with all trial participants, outcome assessors (research staff and care providers), investigators, and trials statistician and data analysts being unable to determine the allocated trial arm for any trial participant or identify trial participants who are on the same trial regimen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- MM 30mg; then MMS 45mg; then MMS 60mg (Experimental): Participants first receive MMS with 30 mg for one month, then MMS with 45 mg of iron for one month, then MMS with 60 mg of iron for one month
  Interventions: Dietary Supplement: Multiple Micronutrient Supplements with 30 mg of elemental iron; Dietary Supplement: Multiple Micronutrient Supplements with 45 mg of elemental iron; Dietary Supplement: Multiple Micronutrient Supplements with 60 mg of elemental iron
- MM 30mg; then MMS 60mg; then MMS 45mg (Experimental): Participants first receive MMS with 30mg for one month, then MMS with 60mg of iron for one month, then MMS with 45 mg of iron for one month
  Interventions: Dietary Supplement: Multiple Micronutrient Supplements with 30 mg of elemental iron; Dietary Supplement: Multiple Micronutrient Supplements with 45 mg of elemental iron; Dietary Supplement: Multiple Micronutrient Supplements with 60 mg of elemental iron
- MM 45mg; then MMS 30mg; then MMS 60mg (Experimental): Participants first receive MMS with 45 mg for one month, then MMS with 30 mg of iron for one month, then MMS with 60 mg of iron for one month
  Interventions: Dietary Supplement: Multiple Micronutrient Supplements with 30 mg of elemental iron; Dietary Supplement: Multiple Micronutrient Supplements with 45 mg of elemental iron; Dietary Supplement: Multiple Micronutrient Supplements with 60 mg of elemental iron
- MM 45 mg; then MMS 60mg; then MMS 30mg (Experimental): Participants first receive MMS with 45 mg for one month, then MMS with 60 mg of iron for one month, then MMS with 30 mg of iron for one month
  Interventions: Dietary Supplement: Multiple Micronutrient Supplements with 30 mg of elemental iron; Dietary Supplement: Multiple Micronutrient Supplements with 45 mg of elemental iron; Dietary Supplement: Multiple Micronutrient Supplements with 60 mg of elemental iron
- MM 60mg; then MMS 30mg; then MMS 45mg (Experimental): Participants first receive MMS with 60 mg for one month, then MMS with 30 mg of iron for one month, then MMS with 45 mg of iron for one month
  Interventions: Dietary Supplement: Multiple Micronutrient Supplements with 30 mg of elemental iron; Dietary Supplement: Multiple Micronutrient Supplements with 45 mg of elemental iron; Dietary Supplement: Multiple Micronutrient Supplements with 60 mg of elemental iron
- MM 60mg; then MMS 45mg; then MMS 30mg (Experimental): Participants first receive MMS with 60 mg for one month, then MMS with 45 mg of iron for one month, then MMS with 30 mg of iron for one month
  Interventions: Dietary Supplement: Multiple Micronutrient Supplements with 30 mg of elemental iron; Dietary Supplement: Multiple Micronutrient Supplements with 45 mg of elemental iron; Dietary Supplement: Multiple Micronutrient Supplements with 60 mg of elemental iron

INTERVENTIONS:
Dietary Supplement: Multiple Micronutrient Supplements with 30 mg of elemental iron — MMS with 30 mg iron is the active comparator group. The standard UNIMMAP MMS formulation includes 30 mg of iron which will be taken orally once daily for one month.
Dietary Supplement: Multiple Micronutrient Supplements with 45 mg of elemental iron — MMS with 45 mg iron is an intervention group. MMS with 45 mg of iron plus standard UNIMMAP formulation for other 14 micronutrients will be taken orally once daily for one month.
Dietary Supplement: Multiple Micronutrient Supplements with 60 mg of elemental iron — MMS with 60 mg iron is an intervention group. MMS with 60 mg of iron plus standard UNIMMAP formulation for other 14 micronutrients will be taken orally once daily for one month.

SUMMARY:
This is an individually randomized cross-over trial to assess acceptability, preference, and perceived side effects of MMS formulations with 30 mg, 45 mg and 60 mg of iron.

ELIGIBILITY:
Inclusion Criteria:

* Attending first ANC visit at the study clinic
* Pregnant women ≤ 15 weeks of gestation
* Aged ≥ 18 years
* Intending to stay in Dar es Salaam for the duration of study
* Provides informed consent

Exclusion Criteria:

* Severe anemia (defined as Hb <8.5 g/dL per Tanzania standard of care)
* Sickle cell disease (SS,SC, CC genotype) as tested by HemoTypeSC
* Concurrent participation in other nutritional supplementation trial
* Pregnant women with disability or condition which would impair their ability to provide informed consent and complete study procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2026-01-23 (Actual); Study Completion 2026-04-24 (Estimated)

PRIMARY OUTCOMES:
Acceptability of MMS formulations | At one month of taking each regimen, up to 3 months
  Participant reported acceptability of each MMS formulation using Likert scales ranging from 1 (disliked a lot) to 5 (liked a lot).

SECONDARY OUTCOMES:
Most preferred MMS formulation | At three months (after taking all three regimens)
  Participant's reported preference for MMS formulations with 30 mg, 45 mg, or 60 mg of iron by asking which supplement participant likes the best.
Least preferred MMS formulation | At three months (after taking all three regimens)
  Participant's reported preference for MMS formulations with 30 mg, 45 mg, or 60 mg of iron by asking which supplement participant likes the least.
Identification of MMS iron dosage | At three months (after taking all three regimens)
  Percentage of participants that correctly identify their iron dose treatment order
Side effects of MMS formulations | At one month of taking each regimen, up to 3 months
  The percentage of patients experiencing any side effect (diarrhea, heartburn, constipation, vomiting, nausea, leg cramps, lower back/pelvic pain) during each intervention period
Adherence | At one month of taking each regimen, up to 3 months
  The percentage of days a participant takes a MMS pill out of the total number of days in the intervention period

OTHER OUTCOMES:
Diarrhea | At one month of taking each regimen, up to 3 months
  The percentage of patients with self-reported diarrhea symptoms during each intervention period
Heartburn | At one month of taking each regimen, up to 3 months
  The percentage of patients with self-reported heartburn symptoms during each intervention period
Constipation | At one month of taking each regimen, up to 3 months
  The percentage of patients with self-reported constipation symptoms during each intervention period
Vomiting | At one month of taking each regimen, up to 3 months
  The percentage of patients with self-reported vomiting during each intervention period
Nausea | At one month of taking each regimen, up to 3 months
  The percentage of patients with self-reported nausea symptoms during each intervention period
Leg cramps | At one month of taking each regimen, up to 3 months
  The percentage of patients with self-reported leg cramp symptoms during each intervention period
Lower back/pelvic pain | At one month of taking each regimen, up to 3 months
  The percentage of patients with self-reported lower back/pelvic painsymptoms during each intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Blair Wylie, MD, MPH, Principal Investigator — Columbia University; Honorati Masanja, PhD, Principal Investigator — Ifakara Health Institute; Alfa Muhihi, PhD, Principal Investigator — Africa Academy for Public Health; Andreas Pembe, MD, MMed, PhD, FCOG, Principal Investigator — Muhimbili University of Health and Allied Sciences; Emily R Smith, ScD, MPH, Principal Investigator — The George Washington University; Christopher R Sudfeld, ScD, ScM, Principal Investigator — Harvard University
Locations (1):
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania